CLINICAL TRIAL: NCT00609960
Title: Clowns as Treatment for Preoperative Anxietyin Children- a Randomized Controlled Trial
Brief Title: Clowns as Treatment for Preoperative Anxiety in Children: A Randomized Controlled Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sheba Medical Center (Other Government)
Responsible Party: Ilan Keidan MD, Director pediatric anesthesia, Sheba Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: SHEBA-05-3739-IK-CTIL
Record Dates: First submitted 2008-01-24; First posted 2008-02-07 (Estimated); Last update posted 2008-02-07 (Estimated); Status verified 2008-01

CONDITIONS: Pre Operative Anxiety
Keywords: children anesthesia anxiety clowns
MeSH Terms: interventions — Midazolam

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (No Intervention): no medication or clowns present during the preopertaive phase
- 2 (Active Comparator): midazolam a anxiolytic drug was given in the preoperative phase
  Interventions: Drug: midazolam
- 3 (Active Comparator): clowns where present during the preoperative phase
  Interventions: Behavioral: clowns present

INTERVENTIONS:
Behavioral: clowns present — clowns present during the proccess of induction of anesthesia
  Arms: 3
Drug: midazolam — midazolam
  Arms: 2

SUMMARY:
This study wants to test the hypothesis that trained clowns can reduce anxiety in children undergoing general anesthesia. We will compare the effect of the clowns to the commonly used anti-anxiety medication we commonly use

DETAILED DESCRIPTION:
The perioperative environment, often anxiety-provoking for adults, may be quite frightening for children. The detrimental effects of preoperative anxiety are not confined to the preoperative period. Anxiety during induction of anesthesia is correlated with increased distress early in the postoperative period, (Holms Knud, Kain) and maladaptive behavior will follow for the first 2 weeks following surgery in up to 54% of children.

Many preoperative systems allow parental, pharmacologic, and anticipatory interventions to facilitate a relaxed perioperative environment for children. Unfortunately, scheduling conflicts, side effects, and limited resources conspire to limit their usefulness. For example, only 10% of respondents in a recent survey used parental presence during induction of anesthesia (PPIA) for a majority of their patients. This may be due to the belief by some that parental anxiety may in fact increase children's anxiety. (Bevans) According to the same survey, only 50% of children undergoing surgery receive sedating premedication. (Kain). Distraction techniques, such as the use of toys or video games, may also decrease perioperative anxiety, however their effectiveness during induction of anesthesia is not well characterized. The efficacy of toys and video games is somewhat dependent upon the child reaching certain developmental milestones. Anesthesiologists continue to search for an easy and comprehensive method for anxiety reduction in the pediatric surgical population. We propose that specially trained professional clowns may allay preoperative anxiety and result in a smooth anesthetic induction.

ELIGIBILITY:
Inclusion Criteria:

* ASA I and II
* Children aged 2-8 years

Exclusion Criteria:

* Previous surgery
* ASA > II
* Parents' refusal

Ages: 2 Years to 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 65 (Actual)
Dates: Start 2006-01; Primary Completion 2007-01 (Actual); Study Completion 2007-01 (Actual)

PRIMARY OUTCOMES:
anxiety level | waiting area and enterance to OR -1 hour

CONTACTS AND LOCATIONS:
Overall Officials: Ilan Keidan, MD, Principal Investigator — Sheba Medical Center
Locations (1):
- Sheba Medical Center, Tel Litwinsky, Ramat Gan, Israel